CLINICAL TRIAL: NCT04638491
Title: Phase 1, Single-arm, Open-label, Dose Escalating and Expansion Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic and Preliminary Efficacy of Lurbinectedin (PM01183) for Injection in Patients With Advanced Solid Tumors
Brief Title: Safety Tolerability Pharmacokinetic and Preliminary Efficacy in Chinese Advanced Solid Tumors Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY01017/CT-CHN-101
Record Dates: First submitted 2020-11-05; First posted 2020-11-20 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumor
Keywords: Lurbinectedin(PM01183) for injection
MeSH Terms: interventions — PM 01183; Injections

STUDY DESIGN:
Intervention Model Description: Lurbinectedin for injection(PM01183)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single-arm (Experimental): PM01183-Dose Escalation
  Interventions: Drug: Lurbinectedin for injection

INTERVENTIONS:
Drug: Lurbinectedin for injection — On the first day of each cycle, patients with advancedsolid tumors or small cell lung cancer were treated with Lurbinectedin for injection
  Other Names: PM01183

SUMMARY:
Phase 1, single-arm, open-label, dose escalating and expansion clinical trial to evaluate the safety, tolerability, pharmacokinetic and preliminary efficacy of Lurbinectedin (PM01183) for injection in patients with advanced solid tumors

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of PM01183 as a single agent, and to identify the dose limiting toxicities (DLTs), determine the recommended dose (RD) in Chinese advanced solid tumors patients

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary written informed consent of the patient.
* 2. Age≥18 years.
* 3. Escalating stage: Patients with histologically/cytologically confirmed diagnosis of advanced solid tumors refractory to standard therapy or for whom refuses or cannot tolerate standard treatment or no standard therapy exist (no more than three prior regimens for advanced or unresectable disease).
* 4. Expansion stage: Patients with histologically confirmed diagnosis of advanced or unresectable SCLC who had failure to one prior platinum -containing line.
* 5. Measurable disease as defined by the RECIST v.1.1.
* 6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
* 7. Life expectancy ≥3 months.
* 8. Adequate bone marrow, renal, hepatic, and metabolic function as follows: Platelet count ≥ 100 x 109/l, Hemoglobin ≥ 90 g/l, absolute neutrophil count (ANC) ≥ 2.0 x 109/l; Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 3.0 x upper limit of normal (ULN), ≤ 5.0 x ULN if presence of liver metastases; Alkaline phosphatase ≤ 5.0 x ULN ; Total bilirubin ≤ 1.5 x ULN, and direct bilirubin ≤1 x ULN ; Serum creatinine ≤ 1.5 x ULN or Calculated creatinine clearance: ≥ 30 ml/min (calculated using the Cockcroft and Gault formula); Creatine phosphokinase (CPK) ≤ 2.5 x ULN; Albumin ≥ 3 g/dl.
* 9. Recovery to grade ≤ 1 according to the NCI-CTCAE v.5.0, of any ongoing adverse event derived from previous treatment ( with the exception of grade 2 alopecia and non-painful peripheral sensory neuropathy ).
* 10. Women of childbearing potential must have a negative serum pregnancy test before study entry. Women of childbearing potential must agree to use a medically acceptable method of contraception throughout the treatment period and for 6 months after discontinuation of treatment. Male patients (female partners is of childbearing potential ) take effective contraceptive measures throughout the treatment period and for 4 months after discontinuation of treatment.

Exclusion Criteria:

* 1. Prior treatment with trabectedin.
* 2. Patients with brain metastases, a history of spinal cord compression, or meningeal metastases.
* 3. Suspected or confirmed disease bone marrow involved.
* 4. Bone metastases, obstructive atelectasis, superior vena cava syndrome patients with local symptoms that may require radiotherapy/surgery/endoscopic treatment/interventional intervention; patients with suspected or confirmed pulmonary embolism; uncontrollable large amounts of pleural fluid, ascites and pericardial effusion.
* 5. Patients who received other recent antitumor therapies ( with respect to study treatment start ) : Less than three weeks since the last chemotherapy-containing regimen (six weeks in case of nitrosoureas, mitomycin C ).

Less than four weeks since the last monoclonal antibody-containing therapy or radiotherapy (RT) dose >30 Gy.

Less than two weeks since the last any other biological/investigational anticancer therapy or palliative radiotherapy ( total dose ≤30 Gy).

* 6. Concomitant diseases/conditions: History (during the last year) or presence of any of the following: unstable angina, myocardial infarction, New York Heart Association (NYHA) Class II or greater congestive heart failure (CHF), or clinically significant valvular heart disease; History of stroke within 1 year (including ischemic stroke, hemorrhagic stroke); Patients with uncontrolled hypertension (systolic blood pressure greater than 160 mmHg and/or diastolic blood pressure greater than 100 mmHg); History of hypertensive crisis or hypertensive encephalopathy; Severe arrhythmia requiring ongoing pharmacological treatment; Positive tests for Hepatitis B surface antigen (HBsAg) and the peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) titer test is ≥1×103 copies/mL; if the HBsAg is positive, and the peripheral blood HBV DNA titer test is <1×103 copies/ml and in the Investigator's judgment, the patient is under a stable stage of chronic hepatitis B and does not increase the risk of the patient, then the patient is eligible for selection; HCV antibody positive or HIV antibody positive; Active uncontrolled infection requiring ongoing medical treatment within two weeks prior to treatment start.

Evidence of bleeding diathesis or significant coagulopathy; Prior or concurrent invasive malignancy other than the primary study indication within 5 years prior to treatment start, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and ductal carcinoma in situ after radical resection； Any other major illness that, in the Investigator's judgment, not suitable for inclusion in this study.

* 7. History of previous bone marrow and/or stem cell transplantation.
* 8. Prior medication requirements: Patients who have used strong inducers or inhibitors of cytochrome P450 3A4 enzyme (CYP3A4) within 2 weeks or 5 half-lives ( whichever is longer ) prior to treatment start; Prophylaxis or treatment for non-febrile neutropenia with G-CSF within two weeks prior to treatment start; Patients who have used erythropoietin and derivatives within 3 weeks prior to treatment start; Patients who have used blood transfusions within 2 weeks prior to treatment start.
* 9. Patients who may need to receive other systemic anti-tumor or radical treatments for local target/non-target lesions during the study period;
* 10. Known history of psychotropic drug, alcohol or drug abuse;
* 11. Known to be allergic to any component of the investigational drug;
* 12. Pregnant or breastfeeding women, or women of childbearing potential have a positive blood pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | From date of first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months(each cycle is 21 days)
  The number and percentage of subjects with significant remission (CR + PR) were calculated, and the 95% confidence interval of the percentage was calculat

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | From date of first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months(each cycle is 21 days)
  The number and percentage of subjects with disease control (CR+PR+SD) were calculated, and the 95% confidence interval of the percentage was calculated
Progression Free Survival(PFS) | From date of first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months(each cycle is 21 days)
  Survival analysis (Kaplan Meier method) was used to estimate the median dor and its 95% confidence interval (CI), and the K-M curve was drawn
Overall Survival(OS) | From date of first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months(each cycle is 21 days)
  Survival analysis (Kaplan Meier method) was used to estimate the median dor and its 95% confidence interval (CI), and the K-M curve was drawn
Duration of remission (DOR) | From date of first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months(each cycle is 21 days)
  Survival analysis (Kaplan Meier method) was used to estimate the median dor and its 95% confidence interval (CI), and the K-M curve was drawn

CONTACTS AND LOCATIONS:
Overall Officials: cheng ying, Doctor, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (1):
- Jilin Provincial Tumor Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng Y, Wu C, Wu L, Zhao J, Zhao Y, Chen L, Xin Y, Zhang L, Pan P, Li X, Li J, Dong X, Tang K, Gao E, Yu F. A pivotal bridging study of lurbinectedin as second-line therapy in Chinese patients with small cell lung cancer. Sci Rep. 2024 Feb 13;14(1):3598. doi: 10.1038/s41598-024-54223-5. PMID 38351146